CLINICAL TRIAL: NCT02965794
Title: Descriptive Study to Evaluate the Care Process and the Quality of Care for Adult Cancer Patients Who Are Admitted for Colorectal Cancer Surgery.
Brief Title: Care Pathways for Colorectal Cancer Surgery
Acronym: CP4GICAN
Status: Completed | Type: Observational
Sponsor: European Pathway Association (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Principal Investigator, Dr. Kris Vanhaecht, Professor in Healthcare Quality Management, European Pathway Association
Other Study IDs: CP4NutriGICAN2014
Record Dates: First submitted 2014-08-04; First posted 2016-11-17 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2019-01

CONDITIONS: Cancer
Keywords: surgery; bowel; rectum; cancer; nutrition
MeSH Terms: conditions — Neoplasms | interventions — Critical Pathways

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Usual care: quality of care will be measured in the participating hospitals, using a retrospective patient record analysis
- Care Pathway: Care pathways for colorectal cancer
  Interventions: Other: Care pathways for colorectal cancer

INTERVENTIONS:
Other: Care pathways for colorectal cancer — development of a care pathway for this patient group
  Other Names: care pathway; clinical pathway; critical pathway
  Groups: Care Pathway

SUMMARY:
EVALUATE THE CARE PROCESS AND THE QUALITY OF CARE FOR ADULT CANCER PATIENTS WHO ARE ADMITTED FOR COLORECTAL SURGERY

DETAILED DESCRIPTION:
This descriptive study uses an interrupted time series approach combining a retrospective with a prospective multicenter design to evaluate the current state of the care process for adult colorectal cancer patients who are admitted for surgery. This study will give attention to evidence based key interventions, follow-up and interprofessional teamwork necessary to provide appropriate care. In 4 countries (Belgium, Germany, France and The Netherlands) 3 hospitals will participate (total number of hospitals is 12). They will perform a clinical audit of the actual organization of the care process, and a team audit on the level of interprofessional teamwork. Each team will develop and implement a quality improvement initiative based on the concept of care pathways, the findings from the audit and the available evidence, and will measure the effect of their improvement strategy.

ELIGIBILITY:
Inclusion Criteria:

1. All consecutive scheduled admissions starting September 2, 2013;
2. Minimum age of 18 years;
3. Elective admission for colorectal cancer surgery

Exclusion Criteria:

1. Emergency (not planned) admission for colorectal cancer surgery;
2. Patients with severe dementia (DSM IV) or severe concomitant disease that may affect very short-term outcome (life expectancy less than 3 months) and hence influence deviations from standard acute care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults undergoing surgery for colorectal cancer
Sampling Method: Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2014-10; Primary Completion 2018-12 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Length of stay | through study completion, an average of 4 months
  Number of days in hospital

SECONDARY OUTCOMES:
Time to return to normal diet | through study completion, an average of 4 months
  number of days in between surgery and day of normal diet

CONTACTS AND LOCATIONS:
Overall Officials: Kris Vanhaecht, PhD, Principal Investigator — KU Leuven
Locations (1):
- KULeuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Zelm R, Coeckelberghs E, Sermeus W, Wolthuis A, Bruyneel L, Panella M, Vanhaecht K. A mixed methods multiple case study to evaluate the implementation of a care pathway for colorectal cancer surgery using extended normalization process theory. BMC Health Serv Res. 2021 Jan 4;21(1):11. doi: 10.1186/s12913-020-06011-w. PMID 33397382